CLINICAL TRIAL: NCT01390948
Title: A Phase II Open-Label, Randomized, Multi-Centre Comparative Study Of Bevacizumab-Based Therapy In Paediatric Patients With Newly Diagnosed Supratentorial, Infratentorial Cerebellar, or Peduncular High-Grade Glioma
Brief Title: A Study of Bevacizumab (Avastin) in Combination With Temozolomide (TMZ) and Radiotherapy in Paediatric and Adolescent Participants With High-Grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO25041; 2010-022189-28 (EudraCT Number); ITCC-019 (Other: Innovative Therapies for Children with Cancer Consortium (ITCC)); HGG-01 (Other: SIOP-E-Brain Tumour Group)
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Results first posted 2017-08-04 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: High Grade Glioma
MeSH Terms: conditions — Glioma | interventions — Bevacizumab; Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bevacizumab + TMZ Young Patient Cohort (YPC) (Experimental): Participants aged greater than or equal to (>/=) 6 months and less than (<) 3 years will receive 10 milligrams per kilogram (mg/kg) Bevacizumab every 2 weeks and 150 to 200 milligrams per meter squared (mg/m^2) of TMZ daily on Days 1-5 of each cycle. TMZ will be given at a dose of 150 mg/m^2 on Days 1-5 of cycle 1 and then escalated to 200 mg/m^2 on days 1-5 from cycle 2 onwards depending on the tolerance during the 1st cycle.
  Interventions: Drug: Bevacizumab; Drug: Temozolomide (TMZ)
- Main Cohort: Chemoradiation + Bevacizumab + TMZ (Experimental): Participants will receive a total dose of 54 Grey (Gy) units delivered in 30 daily fractions of 1.8 Gy over 6 weeks with 75 mg/m^2 TMZ daily for up to 49 days followed by a treatment break of approximately 4 weeks. The treatment break will be followed by an adjuvant treatment phase where participants will receive 150 to 200 mg/m^2 of TMZ daily on Days 1-5 of each cycle. TMZ will be given at a dose of 150 mg/m^2 on Days 1-5 of cycle 1 and then escalated to 200 mg/m^2 on days 1-5 from cycle 2 onwards depending on the tolerance during the 1st cycle. Bevacizumab will be given concomitantly at a dose of 10 mg/kg every 2 weeks throughout the entire treatment period.
  Interventions: Drug: Bevacizumab; Radiation: Radiotherapy; Drug: Temozolomide (TMZ)
- Main Cohort: Chemoradiation + TMZ (Active Comparator): Participants will receive a total dose of 54 Gy units delivered in 30 daily fractions of 1.8 Gy over 6 weeks with 75 mg/m^2 TMZ daily for up to 49 days followed by a treatment break of approximately 4 weeks. The treatment break will be followed by an adjuvant treatment phase where participants will receive 150 to 200 mg/m^2 of TMZ daily on Days 1-5 of each cycle. TMZ will be given at a dose of 150 mg/m^2 on Days 1-5 of cycle 1 and then escalated to 200 mg/m^2 on days 1-5 from cycle 2 onwards depending on the tolerance during the 1st cycle.
  Interventions: Radiation: Radiotherapy; Drug: Temozolomide (TMZ)

INTERVENTIONS:
Drug: Bevacizumab — 10 milligrams per kilogram every 2 weeks during the study for up to 12 cycles, each cycle length of 28 days
  Other Names: Avastin
  Arms: Bevacizumab + TMZ Young Patient Cohort (YPC); Main Cohort: Chemoradiation + Bevacizumab + TMZ
Radiation: Radiotherapy — Total dose of 54 Grey (Gy) units delivered in 30 daily fractions of 1.8 Gy over 6 weeks during the chemoradiation phase.
  Arms: Main Cohort: Chemoradiation + Bevacizumab + TMZ; Main Cohort: Chemoradiation + TMZ
Drug: Temozolomide (TMZ) — 75 milligrams per square meter (mg/m^2) daily continuous starting concomitantly with the first radiation fraction and ending with the last radiation fraction for a maximum number of treatment days = 49 days. During the TMZ adjuvant treatment phase and for participants from YPC: TMZ (150 to 200 mg/m^2/day) x 12 cycles, 1st cycle 150 mg/m^2/days 1-5, escalated to 200 mg/m^2 on Days 1-5 from Cycle 2 onwards depending on the tolerance during the 1st cycle. Cycle length = 28 days.

SUMMARY:
This randomized, open-label, multicenter, 2-arm study will investigate the efficacy, safety, tolerability and pharmacokinetics of bevacizumab when added to postoperative radiotherapy with concomitant and adjuvant TMZ as compared to postoperative radiotherapy with concomitant and adjuvant TMZ alone in paediatric participants with newly diagnosed histologically confirmed World Health Organization (WHO) Grade III or IV localized supratentorial or infratentorial cerebellar or peduncular high grade glioma (HGG). Participants will be randomly assigned to one of two treatment arms.

Upon approval by the Health Authorities/Ethics Committees in the participating countries, an additional young participant cohort (YPC) (children >/= 6 months and < 3 years of age with progressive or relapsed metastatic or localized, supra- or infratentorial, non-brain stem WHO Grade III or IV HGG) was included in the study. Children in the YPC will receive bevacizumab and TMZ without radiation therapy. The anticipated time on study treatment is over 1 year.

ELIGIBILITY:
Inclusion Criteria - Main cohort :

* Paediatric participants, aged >= 3 years and < 18 years
* Written informed consent obtained from the participant/parents or legally acceptable representative
* Newly diagnosed localised, supratentorial or infratentorial cerebellar or peduncular, WHO Grade III or IV gliomas
* Local histological diagnosis confirmed by a designated central reference neuropathologist
* Availability of the baseline magnetic resonance imaging (MRI) performed according to imaging guidelines
* Able to commence trial treatment not before 4 weeks after cranial surgery and no later than 6 weeks following the last major surgery
* Adequate bone marrow, coagulation, liver, and renal function

Young Participant Cohort

* Written informed consent obtained from parents or legal representative
* Age at enrollment: from >= 6 months to < 3 years of age
* Progressive or relapsed metastatic or localised, supra- or infratentorial, non-brain stem WHO Grade III or IV glioma (local pathology confirmation made either at initial diagnosis or at relapse)
* Availability of a baseline MRI performed according to imaging guidelines
* Adequate organ function (bone marrow, coagulation, liver, kidney)

Exclusion Criteria - Main cohort:

* Metastatic HGG defined as evidence of neuraxis dissemination by MRI or positive cerebrospinal fluid (CSF) cytology
* WHO-defined Gliomatosis cerebri (multifocal HGG)
* Any disease or condition that contraindicates the use of the study medication/treatment or places the patient at an unacceptable risk of experiencing treatment-related complications
* Radiological evidence of surgically related intracranial bleeding
* Prior diagnosis of a malignancy and disease-free for 5 years
* Prior systemic anti-cancer therapy
* Previous cranial irradiation

Young Participant Cohort

* WHO-defined Gliomatosis cerebri (multifocal HGG)
* Newly diagnosed HGG below the age of 3 years
* Relapsed HGG below the age of 6 months or above the age of 3 years regardless of the age at first onset
* Indication for concomitant cranial irradiation, regardless of age
* Any disease or condition that contraindicates the use of the study medication/treatment or places the child at an unacceptable risk of experiencing treatment-related complications
* Any specific contraindication to MRI

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Actual)
Dates: Start 2011-10-18 (Actual); Primary Completion 2016-02-05 (Actual); Study Completion 2020-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (53):
- Australia (2):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Lady Cilento Children's Hospital; Oncology Services Group, Level 12b, South Brisbane, Queensland
- Austria (2):
  - Kepler Universitätskliniken GmbH - Med Campus IV., Linz
  - Medizinische Universität Wien, Vienna
- UZ Leuven Gasthuisberg, Leuven, Belgium
- Canada (2):
  - Alberta Children'S Hospital, Calgary, Alberta
  - Hospital For Sick Children, Toronto, Ontario
- Czechia (2):
  - Fakultni nemocnice Brno; 2. detska klinika, pracoviste Detska nemocnice, Brno
  - Fakultni Nemocnice V Motole, S.P., Prague
- Denmark (2):
  - Skejby Sygehus - Aarhus University Hospital; CF Center, Børneafdeling A, Aarhus N
  - Rigshospitalet; Onkologisk Klinik, København Ø
- France (14):
  - Centre Hospitalier d'Angers; Service de cancérologie pédiatrique, Angers
  - CHU ESTAING; Centre Regional de Cancérologie et Thérapie Cellulaire Pédiatrique (CRCTCP), Clermont-Ferrand
  - Centre Oscar Lambret; Service de Pediatrie, Lille
  - Centre Leon Berard, Lyon
  - Hopital Timone Enfants; Onco Pediatrie, Marseille
  - Hopital Lenval; Service Hématologie Infantile, Nice
  - Institut Curie - Centre de Lutte Contre le Cancer (CLCC) de Paris; Service d Oncologie Pediatrique, Paris
  - CHRU de Rennes - Hôpital Sud- Service d'Hématologie Pédiatrique, Rennes
  - Hopital Nord;Consult Pediatrie, Saint-Priest-en-Jarez
  - Hôpital Hautepierre, Strasbourg
  - Hopital Des Enfants; Service d Hemato-Oncologie, Toulouse
  - CHRU de Tours - Centre de Pédiatrie Clocheville; Service d'Oncopédiatrie, Tours
  - Hopital Brabois Enfants, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy; Service Pediatrique, Villejuif
- Semmelweis University, 2nd Dept of Pediatrics Neurooncology Unit, Budapest, Hungary
- Italy (4):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpigh, Bologna, Emilia-Romagna
  - Istituto Giannina Gaslini-Ospedale Pediatrico IRCCS; U.O.S. Neuroncologia, Genoa, Liguria
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Azienda Ospedaliera di Padova, Padua, Veneto
- Netherlands (2):
  - UMC St Radboud, Nijmegen
  - Erasmus Mc/Sophia's Childrens Hospital; Dept. of Pediatric Oncology, Rotterdam
- Instytut Pomnik-Centrum Zdrowia Dziecka; Klinika Onkologii, Warsaw, Poland
- Spain (3):
  - Hospital Sant Joan De Deu, Esplugues de Llobregas, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Fe, Valencia
- Sweden (4):
  - Sahlgrenska Universitetssjukhuset, Östra Sjukhus; Drottning Silvias Barnsjukhus, Gothenburg
  - Universitetssjukhuset Linköping; Barn och Ungdomskliniken, Linköping
  - Skånes Universitetssjukhus, Lund
  - Karolinska Universitetssjukhuset, Solna; Astrid Lindgrens Barnsjukhus, Barcanceravdelningen, Solna
- United Kingdom (13):
  - Birmingham Childrens Hospital; Oncology Dept, Birmingham
  - Bristol Royal Hospital for Children; Paediatric Haematology, Oncology, BMT, Bristol
  - Addenbrookes Hospital; Paediatric Oncology Ward C2, Cambridge
  - Royal Hospital for Sick Children, Edinburgh
  - Leeds General Infirmary; Ward 35, Leeds
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - University College London NHS Foundation Trust, London
  - Great Ormond Street Hospital; Dept. Of Pediatric Oncology, London
  - Royal Manchester Childrens Hospital, Manchester
  - Newcastle University & The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Queens Medical Centre, Nottingham
  - Southampton General Hospital, Southampton
  - Royal Marsden Hospital; Pediatric Unit, Surrey

REFERENCES:
- [Derived] Rodriguez D, Calmon R, Aliaga ES, Warren D, Warmuth-Metz M, Jones C, Mackay A, Varlet P, Le Deley MC, Hargrave D, Canete A, Massimino M, Azizi AA, Saran F, Zahlmann G, Garcia J, Vassal G, Grill J, Peet A, Dineen RA, Morgan PS, Jaspan T. MRI and Molecular Characterization of Pediatric High-Grade Midline Thalamic Gliomas: The HERBY Phase II Trial. Radiology. 2022 Jul;304(1):174-182. doi: 10.1148/radiol.211464. Epub 2022 Apr 12. PMID 35412366
- [Derived] Varlet P, Le Teuff G, Le Deley MC, Giangaspero F, Haberler C, Jacques TS, Figarella-Branger D, Pietsch T, Andreiuolo F, Deroulers C, Jaspan T, Jones C, Grill J. WHO grade has no prognostic value in the pediatric high-grade glioma included in the HERBY trial. Neuro Oncol. 2020 Jan 11;22(1):116-127. doi: 10.1093/neuonc/noz142. PMID 31419298
- [Derived] Rodriguez D, Chambers T, Warmuth-Metz M, Aliaga ES, Warren D, Calmon R, Hargrave D, Garcia J, Vassal G, Grill J, Zahlmann G, Morgan PS, Jaspan T. Evaluation of the Implementation of the Response Assessment in Neuro-Oncology Criteria in the HERBY Trial of Pediatric Patients with Newly Diagnosed High-Grade Gliomas. AJNR Am J Neuroradiol. 2019 Mar;40(3):568-575. doi: 10.3174/ajnr.A5982. Epub 2019 Feb 28. PMID 30819765
- [Derived] Mackay A, Burford A, Molinari V, Jones DTW, Izquierdo E, Brouwer-Visser J, Giangaspero F, Haberler C, Pietsch T, Jacques TS, Figarella-Branger D, Rodriguez D, Morgan PS, Raman P, Waanders AJ, Resnick AC, Massimino M, Garre ML, Smith H, Capper D, Pfister SM, Wurdinger T, Tam R, Garcia J, Thakur MD, Vassal G, Grill J, Jaspan T, Varlet P, Jones C. Molecular, Pathological, Radiological, and Immune Profiling of Non-brainstem Pediatric High-Grade Glioma from the HERBY Phase II Randomized Trial. Cancer Cell. 2018 May 14;33(5):829-842.e5. doi: 10.1016/j.ccell.2018.04.004. PMID 29763623
- [Derived] Grill J, Massimino M, Bouffet E, Azizi AA, McCowage G, Canete A, Saran F, Le Deley MC, Varlet P, Morgan PS, Jaspan T, Jones C, Giangaspero F, Smith H, Garcia J, Elze MC, Rousseau RF, Abrey L, Hargrave D, Vassal G. Phase II, Open-Label, Randomized, Multicenter Trial (HERBY) of Bevacizumab in Pediatric Patients With Newly Diagnosed High-Grade Glioma. J Clin Oncol. 2018 Apr 1;36(10):951-958. doi: 10.1200/JCO.2017.76.0611. Epub 2018 Feb 7. PMID 29412784

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Chemoradiation + temozolomide (TMZ) and Chemoradiation + Bevacizumab + TMZ arms: 174 participants were screened; 121 were randomized; 116 received study treatment. Young Patient Cohort: 4 participants were screened; 3 were enrolled and received study treatment (these subjects were not randomized and are not included in efficacy analyses).
Groups:
- Chemoradiation + TMZ: Participants received a total dose of 54 Grey (Gy) units delivered in 30 daily fractions of 1.8 Gy over 6 weeks with 75 milligrams per meter squared (mg/m^2) TMZ daily for up to 49 days followed by a treatment break of approximately 4 weeks. The treatment break was followed by an adjuvant treatment phase where participants received 150 to 200 mg/m^2 of TMZ daily on Days 1-5 of each cycle. TMZ was given at a dose of 150 mg/m^2 on Days 1-5 of cycle 1 and then escalated to 200 mg/m^2 on days 1-5 from cycle 2 onwards depending on the tolerance during the 1st cycle.
- Chemoradiation + Bevacizumab + TMZ: Participants received a total dose of 54 Gy units delivered in 30 daily fractions of 1.8 Gy over 6 weeks with 75 mg/m^2 TMZ daily for up to 49 days followed by a treatment break of approximately 4 weeks. The treatment break was followed by an adjuvant treatment phase where participants received 150 to 200 mg/m^2 of TMZ daily on Days 1-5 of each cycle. TMZ was given at a dose of 150 mg/m^2 on Days 1-5 of cycle 1 and then escalated to 200 mg/m^2 on days 1-5 from cycle 2 onwards depending on the tolerance during the 1st cycle. Bevacizumab was given concomitantly at a dose of 10 milligrams per kilogram (mg/kg) every 2 weeks throughout the entire treatment period.
- Bevacizumab + TMZ Young Patient Cohort (YPC): Participants aged >/= 6 months and < 3 years received 10 mg/kg Bevacizumab every 2 weeks and 150 to 200 mg/m^2 of TMZ daily on Days 1-5 of each cycle. TMZ was given at a dose of 150 mg/m^2 on Days 1-5 of cycle 1 and then escalated to 200 mg/m^2 on days 1-5 from cycle 2 onwards depending on the tolerance during the 1st cycle.
Period: Overall Study
Arm/Group | Chemoradiation + TMZ | Chemoradiation + Bevacizumab + TMZ | Bevacizumab + TMZ Young Patient Cohort (YPC)
Started | 59 | 62 | 3
Treated | 56 | 60 | 3
Completed | 44 | 44 | 2
Not Completed | 15 | 18 | 1
Not completed — End of Study | 1 | 0 | 0
Not completed — Withdrew consent | 2 | 2 | 0
Not completed — Progressive Disease | 2 | 5 | 0
Not completed — Death during follow-up | 10 | 11 | 1

BASELINE CHARACTERISTICS:
Groups:
- Chemoradiation + TMZ: Participants received a total dose of 54 Gy units delivered in 30 daily fractions of 1.8 Gy over 6 weeks with 75 mg/m^2 TMZ daily for up to 49 days followed by a treatment break of approximately 4 weeks. The treatment break was followed by an adjuvant treatment phase where participants received 150 to 200 mg/m^2 of TMZ daily on Days 1-5 of each cycle. TMZ was given at a dose of 150 mg/m^2 on Days 1-5 of cycle 1 and then escalated to 200 mg/m^2 on days 1-5 from cycle 2 onwards depending on the tolerance during the 1st cycle.
- Chemoradiation + Bevacizumab + TMZ: Participants received a total dose of 54 Gy units delivered in 30 daily fractions of 1.8 Gy over 6 weeks with 75 mg/m^2 TMZ daily for up to 49 days followed by a treatment break of approximately 4 weeks. The treatment break was followed by an adjuvant treatment phase where participants received 150 to 200 mg/m^2 of TMZ daily on Days 1-5 of each cycle. TMZ was given at a dose of 150 mg/m^2 on Days 1-5 of cycle 1 and then escalated to 200 mg/m^2 on days 1-5 from cycle 2 onwards depending on the tolerance during the 1st cycle. Bevacizumab was given concomitantly at a dose of 10 mg/kg every 2 weeks throughout the entire treatment period.
- Total: Total of all reporting groups
Arm/Group | Chemoradiation + TMZ | Chemoradiation + Bevacizumab + TMZ | Bevacizumab + TMZ Young Patient Cohort (YPC) | Total
Number analyzed (Participants) | 59 | 62 | 3 | 124
Age, Customized [Count of Participants; unit: Participants]
  < 3 years | 0 | 0 | 3 | 3
  >/= 3 years and < 6 years | 6 | 10 | 0 | 16
  >/= 6 years and < 13 years | 30 | 35 | 0 | 65
  >/= 13 years and < 18 years | 23 | 17 | 0 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 28 | 0 | 51
  Male | 36 | 34 | 3 | 73

OUTCOME MEASURES:

1. Primary Outcome: Event-Free Survival (EFS) as Assessed by the Central Radiology Review Committee (CRRC)
Description: EFS was defined as the time from randomisation to the earliest occurrence of any of the following: tumor progression, tumor recurrence, second primary non- HGG malignancy or death attributable to any cause. Tumor assessments were conducted using magnetic resonance imaging (MRI) and reviewed by the site-independent CRRC using Response Assessment in Neuro-Oncology (RANO) criteria. Tumor progression was defined as clear clinical progression or >/= 25% increase in the sum of the products of perpendicular diameters of the contrast enhancing lesions compared with the smallest tumor measurement obtained either at baseline (if no decrease was observed) or best response and with the subject on stable or increasing doses of corticosteroids. Tumor recurrence was defined as recurrence after tumor was completely resected (no disease present at baseline). EFS was estimated using the Kaplan-Meier method.
Time Frame: From the time of randomization to the date of any defined event (up to 12 months)
Population: Randomized participant population included all randomized participants regardless of whether they received study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemoradiation + TMZ | Chemoradiation + Bevacizumab + TMZ
Number analyzed (Participants) | 59 | 62
months | 11.79 [7.85 to 16.39] | 8.21 [7.75 to 12.68]
Statistical Analysis 1: Comparison: Chemoradiation + TMZ vs Chemoradiation + Bevacizumab + TMZ; Test type: Superiority or Other; p = 0.1292, Log Rank; Hazard Ratio (HR) = 1.44, 95% CI 2-sided [0.90 to 2.30]

2. Secondary Outcome: Overall Survival
Description: Overall Survival was defined as the time of diagnosis to the date of death due to any cause. Overall Survival was estimated using the Kaplan-Meier method.
Time Frame: From the time of randomization to the date of death (up to approximately 60 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemoradiation + TMZ | Chemoradiation + Bevacizumab + TMZ
Number analyzed (Participants) | 59 | 62
months | 20.27 [14.75 to 33.77] | 18.30 [16.20 to 25.69]

3. Secondary Outcome: Percentage of Participants With 1-Year Survival
Description: 1-year survival was estimated using the Kaplan-Meier method.
Time Frame: 1 year after end of treatment
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation + TMZ | Chemoradiation + Bevacizumab + TMZ
Number analyzed (Participants) | 59 | 62
percentage of participants | 67.69 [55.39 to 79.99] | 74.83 [63.79 to 85.87]

4. Secondary Outcome: Percentage of Participants With EFS as Determined by the CRRC at 6 Months
Description: EFS was defined as the time from randomisation to the earliest occurrence of any of the following: tumor progression, tumor recurrence, second primary non- HGG malignancy or death attributable to any cause. Tumor assessments were conducted using MRI and reviewed by the site-independent CRRC using RANO criteria. Tumor progression was defined as clear clinical progression or >/= 25% increase in the sum of the products of perpendicular diameters of the contrast enhancing lesions compared with the smallest tumor measurement obtained either at baseline (if no decrease was observed) or best response and with the subject on stable or increasing doses of corticosteroids. Tumor recurrence was defined as recurrence after tumor was completely resected (no disease present at baseline). EFS was estimated using the Kaplan-Meier method.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation + TMZ | Chemoradiation + Bevacizumab + TMZ
Number analyzed (Participants) | 59 | 62
percentage of participants | 66.46 [52.58 to 77.13] | 68.43 [55.06 to 78.58]

5. Secondary Outcome: Percentage of Participants With EFS as Determined by the CRRC at 1 Year
Description: as for outcome 4
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation + TMZ | Chemoradiation + Bevacizumab + TMZ
Number analyzed (Participants) | 59 | 62
percentage of participants | 48.37 [34.82 to 60.65] | 38.28 [25.79 to 50.64]

6. Secondary Outcome: EFS as Assessed by the Investigator
Description: EFS was defined as the time from randomisation to the earliest occurrence of any of the following: tumor progression, tumor recurrence, second primary non-HGG malignancy or death attributable to any cause. Tumor assessments were conducted using MRI and reviewed by the investigator using RANO criteria. Tumor progression was defined as clear clinical progression or >/= 25% increase in the sum of the products of perpendicular diameters of the contrast enhancing lesions compared with the smallest tumor measurement obtained either at baseline (if no decrease was observed) or best response and with the participant on stable or increasing doses of corticosteroids. Tumor recurrence was defined as recurrence after tumor was completely resected (no disease present at baseline). EFS was estimated using the Kaplan-Meier method.
Time Frame: From the time of randomization to the date of any defined event (up to 12 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemoradiation + TMZ | Chemoradiation + Bevacizumab + TMZ
Number analyzed (Participants) | 59 | 62
months | 11.79 [8.51 to 20.53] | 11.27 [8.11 to 14.49]

7. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a complete response (CR) or partial response (PR) determined on two consecutive occasions >/= 4 weeks apart. Tumor assessments were conducted using MRI and reviewed by the site-independent CRRC using RANO criteria. The following were needed to qualify as CR: complete disappearance of all measurable enhancing lesions sustained for at least 4 weeks by MRI, no steroids above physiological levels, clinical status stable or improved compared to baseline. The following were needed to qualify as PR: ≥ 50% decrease from baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks by MRI, steroid dose not increased compared to baseline, clinical status stable or improved compared to baseline.
Time Frame: From the time of randomization to the date of any defined event (up to 12 months)
Population: Randomized participant population with a measurable lesion at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation + TMZ | Chemoradiation + Bevacizumab + TMZ
Number analyzed (Participants) | 15 | 12
percentage of participants | 40 [19.09 to 66.77] | 41.7 [18.10 to 70.60]

8. Secondary Outcome: Concordance Between Structural Versus Multimodal Imaging for CRRC-Assessed Event-Free Survival
Description: Concordance is presented as the percentage of participants with concordance between assessments. EFS concordance was defined as event Structural assessment and Diffusion Perfusion assessment occurs within 28 days or no event Structural and no Diffusion Perfusion.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Chemoradiation + TMZ | Chemoradiation + Bevacizumab + TMZ
Number analyzed (Participants) | 59 | 62
percentage of participants | 96.6 | 87.1

9. Secondary Outcome: Health Status as Measured by the Health Utility Index (HUI)
Description: HUI is a preference-based, multi-attitude, health-related instrument specifically developed for use with children. HUI consists of eight attributes of health status: vision, hearing, speech, ambulation, dexterity, emotion, cognition and pain. Each attribute had 5 or 6 levels varying from highly impaired to normal. Each of the eight health dimensions was tested separately and a composite score ranging between 1 (perfect health) and 0 (death) was obtained for participants aged 5 years or older.
Time Frame: Baseline, Cycle 6 of the adjuvant phase, end of treatment (approximately 58 weeks post-baseline), and yearly during the follow-up period (maximum 5 years in follow-up)
Population: Randomized participant population aged 5 years or older with a measure at the specified time point. Here, 'n' represents the number of participants with a measure at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chemoradiation + TMZ | Chemoradiation + Bevacizumab + TMZ
Number analyzed (Participants) | 36 | 45
units on a scale
  Baseline | 0.713 (0.317) | 0.730 (0.274)
  Cycle 6, Day 1: number analyzed (Participants) | 30 | 39
  Cycle 6, Day 1 | 0.785 (0.239) | 0.779 (0.232)
  End of Treatment: number analyzed (Participants) | 21 | 21
  End of Treatment | 0.832 (0.216) | 0.820 (0.209)
  Yearly Follow-Up 1: number analyzed (Participants) | 9 | 7
  Yearly Follow-Up 1 | 0.906 (0.110) | 0.926 (0.109)
  Yearly Follow-up 2: number analyzed (Participants) | 9 | 8
  Yearly Follow-up 2 | 0.737 (0.326) | 0.793 (0.219)
  Additional Safety Follow-Up (Visit 2): number analyzed (Participants) | 8 | 10
  Additional Safety Follow-Up (Visit 2) | 0.784 (0.287) | 0.901 (0.147)
  Additional Safety Follow-Up (Visit 4): number analyzed (Participants) | 7 | 6
  Additional Safety Follow-Up (Visit 4) | 0.814 (0.304) | 0.830 (0.143)
  Additional Safety Follow-Up (Visit 6): number analyzed (Participants) | 2 | 2
  Additional Safety Follow-Up (Visit 6) | 1.000 (0.000) | 0.490 (0.537)
  Additional Safety Follow-Up (Visit 8): number analyzed (Participants) | 0 | 1
  Additional Safety Follow-Up (Visit 8) |  | 0.930 (NA) — A single participant was analyzed
  End of Study: number analyzed (Participants) | 3 | 6
  End of Study | 0.647 (0.496) | 0.790 (0.234)

10. Secondary Outcome: Neurological Psychological Function as Measured by the Wechsler Scale
Description: The Wechsler Intelligence Scale for Children version IV (WISC-IV) was used to generate a full scale intelligence quotient (IQ) which represents a child's general intellectual ability. The average IQ score is 100, with lower scores representing lower intellectual ability.
Time Frame: End of treatment (approximately 58 weeks post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chemoradiation + TMZ | Chemoradiation + Bevacizumab + TMZ
Number analyzed (Participants) | 59 | 62
units on a scale | 92.0 (9.8) | 97.0 (18.4)

11. Secondary Outcome: Percentage of Participants Who Completed >/= 90% of Planned Radiotherapy and TMZ Administrations
Time Frame: From the time of randomization of the first participant to the date of clinical cutoff (approximately 60 months)
Population: Safety population included all participants that received study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Chemoradiation + TMZ | Chemoradiation + Bevacizumab + TMZ
Number analyzed (Participants) | 56 | 60
percentage of participants
  Radiotherapy | 94.6 | 98.3
  TMZ | 85.7 | 88.3

12. Secondary Outcome: Percentage of Participants With a Treatment Delay or Discontinuation
Time Frame: From the time of randomization of the first participant to the date of clinical cutoff (approximately 60 months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Chemoradiation + TMZ | Chemoradiation + Bevacizumab + TMZ
Number analyzed (Participants) | 59 | 62
percentage of participants
  AE leading to dose modification/interruption | 60.7 | 71.7
  AE leading to withdrawal from treatment | 5.4 | 21.7

13. Secondary Outcome: Number of Radiotherapy Dose Administrations in the Concurrent Phase
Description: Number of doses were assessed for the concurrent phase, which is the treatment period after the initial treatment phase and including the subsequent treatment break of approximately 4 weeks.
Time Frame: Beginning of the concurrent phase to end of treatment break (10 weeks)
Population: Safety population included all participants that received study drug.
Measure: Median (Full Range); unit: Grays
Arm/Group | Chemoradiation + TMZ | Chemoradiation + Bevacizumab + TMZ
Number analyzed (Participants) | 56 | 60
Grays | 54.0 [4 to 60] | 54.0 [2 to 56]

14. Secondary Outcome: Number of Dose Administrations of TMZ and Bevacizumab in the Concurrent Phase
Description: as for outcome 13
Time Frame: Beginning of the concurrent phase to end of treatment break (10 weeks)
Population: Safety population included all participants that received study drug.
Measure: Median (Full Range); unit: number of dose administrations
Arm/Group | Chemoradiation + TMZ | Chemoradiation + Bevacizumab + TMZ
Number analyzed (Participants) | 56 | 60
number of dose administrations
  TMZ | 42.0 [1 to 50] | 42.0 [3 to 49]
  Bevacizumab | NA [NA to NA] — Bevacizumab not administered for this arm | 6.0 [1 to 10]

15. Secondary Outcome: Percentage of Participants With an Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: From the time of randomization of the first participant to the date of clinical cutoff (approximately 60 months)
Population: Safety population included all participants that received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Chemoradiation + TMZ | Chemoradiation + Bevacizumab + TMZ
Number analyzed (Participants) | 56 | 60
percentage of participants | 100 | 98.3

ADVERSE EVENTS:
Time Frame: From randomization/enrollment of the first participant to date of clinical cut off (approximately 60 months)
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Arm/Group | Chemoradiation + TMZ | Chemoradiation + Bevacizumab + TMZ | Bevacizumab + TMZ Young Patient Cohort (YPC)
Serious Adverse Events (participants affected / at risk) | 27/56 | 35/60 | 0/3
Other Adverse Events (participants affected / at risk) | 56/56 | 60/60 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemoradiation + TMZ (N=56) | Chemoradiation + Bevacizumab + TMZ (N=60) | Bevacizumab + TMZ Young Patient Cohort (YPC) (N=3)
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 5 (6) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
PRECOCIOUS PUBERTY (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0)
EYELID OEDEMA (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
VOMITING (Gastrointestinal disorders) | 3 (3) | 6 (8) | 0 (0)
CATHETER SITE THROMBOSIS (General disorders) | 0 (0) | 1 (1) | 0 (0)
CYST (General disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOTHERMIA (General disorders) | 1 (1) | 0 (0) | 0 (0)
IMPLANT SITE DEHISCENCE (General disorders) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 5 (6) | 12 (17) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
CATHETER SITE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
DEVICE RELATED SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
PSEUDOMONAS INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
SOFT TISSUE INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
TONSILLITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
VASCULAR DEVICE INFECTION (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
HAEMATURIA TRAUMATIC (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
BODY TEMPERATURE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1) | 1 (2) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 2 (4) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0)
ATYPICAL TERATOID/RHABDOID TUMOUR OF CNS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0)
B-CELL TYPE ACUTE LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OSTEOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL CYST (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CEREBROSPINAL FLUID LEAKAGE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (2) | 4 (5) | 0 (0)
HEMIPARESIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
HYDROCEPHALUS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
MONOPLEGIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
PARTIAL SEIZURES (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
POSTERIOR REVERSIBLE ENCEPHALOPATHY SYNDROME (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 7 (12) | 5 (5) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
STATUS EPILEPTICUS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DEVICE OCCLUSION (Product Issues) | 0 (0) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 2 (3) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
BLISTER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemoradiation + TMZ (N=56) | Chemoradiation + Bevacizumab + TMZ (N=60) | Bevacizumab + TMZ Young Patient Cohort (YPC) (N=3)
ANAEMIA (Blood and lymphatic system disorders) | 6 (13) | 5 (9) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 6 (11) | 3 (3) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 3 (4) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 12 (26) | 9 (19) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 8 (20) | 10 (31) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 2 (2) | 3 (3) | 0 (0)
EYE PAIN (Eye disorders) | 4 (4) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 10 (17) | 12 (18) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 6 (7) | 7 (9) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 12 (19) | 18 (29) | 0 (0)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 13 (19) | 14 (22) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 24 (49) | 22 (38) | 0 (0)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0)
VOMITING (Gastrointestinal disorders) | 29 (65) | 36 (89) | 2 (3)
ASTHENIA (General disorders) | 4 (7) | 6 (6) | 0 (0)
FATIGUE (General disorders) | 32 (44) | 26 (36) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 3 (4) | 1 (2) | 0 (0)
PYREXIA (General disorders) | 16 (27) | 15 (31) | 1 (2)
CANDIDA INFECTION (Infections and infestations) | 2 (4) | 0 (0) | 1 (1)
CONJUNCTIVITIS (Infections and infestations) | 5 (5) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
INFLUENZA (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 6 (6) | 10 (10) | 0 (0)
OTITIS MEDIA ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PHARYNGITIS (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 9 (10) | 8 (9) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 (7) | 3 (6) | 2 (4)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
RADIATION INJURY (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 4 (4) | 5 (5) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 6 (6) | 3 (3) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 (3) | 1 (1) | 0 (0)
HEART RATE INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 17 (32) | 16 (29) | 1 (1)
NEUTROPHIL COUNT INCREASED (Investigations) | 3 (3) | 1 (1) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 19 (46) | 18 (42) | 1 (2)
WEIGHT DECREASED (Investigations) | 3 (3) | 6 (8) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 14 (28) | 16 (32) | 1 (1)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 4 (5) | 2 (2) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 21 (28) | 17 (22) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (6) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (3) | 1 (1)
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 2 (2) | 3 (5) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 32 (66) | 34 (63) | 0 (0)
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 4 (5) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 5 (10) | 2 (2) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 3 (5) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 2 (2) | 5 (6) | 0 (0)
INSOMNIA (Psychiatric disorders) | 7 (9) | 2 (2) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 15 (27) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 12 (17) | 19 (30) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 12 (19) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 5 (11) | 7 (8) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 34 (34) | 19 (20) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (9) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (6) | 0 (0)
PURPURA (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (10) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (4) | 11 (17) | 2 (2)
SKIN STRIAE (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 5 (8) | 8 (10) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 7 (10) | 1 (2)
HYPOTENSION (Vascular disorders) | 2 (2) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.